CLINICAL TRIAL: NCT01379547
Title: Procalcitonin to Shorten Antibiotics Duration in ICU Patients- A China, Hong-Kong, Taiwan Multicenter Trial
Brief Title: Procalcitonin to Shorten Antibiotics Duration in ICU Patients
Acronym: ProShort
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other); Ruijin Hospital (Other); Shanghai Jiao Tong University School of Medicine (Other); Chongqing Medical University (Other); Tianjin Medical University General Hospital (Other); Chinese PLA General Hospital (Other); Xinjiang Medical University (Other); Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201101079RB
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Sepsis
Keywords: Procalcitonin; sepsis; ICU; antibiotic; antibiotic duration; Antibiotic treatment duration
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Treatment (Active Comparator): Patients who will be randomized to arm 1 will receive antibiotic therapy with a duration based on conventional practice
  Interventions: Behavioral: Conventional treatment
- procalcitonin-guided antibiotics treatment (Experimental): Patients who will be randomized to arm 2 will receive antibiotics therapy with a duration based on procalcitonin-guided algorithm.
  Interventions: Behavioral: Procalcitonin guided antibiotics treatment algorithm

INTERVENTIONS:
Behavioral: Procalcitonin guided antibiotics treatment algorithm — Patients who will be randomized to arm 2 will receive antibiotics therapy with a duration based on procalcitonin measurement on day 5, 7 and 9.
  Arms: procalcitonin-guided antibiotics treatment
Behavioral: Conventional treatment — Patients who will be randomized to arm 1 will receive antibiotic therapy with a duration based on conventional practice.
  Arms: Conventional Treatment

SUMMARY:
The trial is aimed to show that implementation of a procalcitonin-guided antibiotics algorithm may result in shortened antibiotics course in ICU sepsis patients without inferior outcome as compared to the conventional therapy

DETAILED DESCRIPTION:
The duration of antibiotic therapy in patients with sepsis is largely empirical. An extended treatment course for up to two weeks is a common practice for patients with sepsis in the ICU, despite lack of evidence for this duration of therapy.

Procalcitonin (PCT) is a new biomarker that has high negative predictive value for systemic bacterial infection. The purpose of this trial is to evaluate whether serial PCT measurements can shorten antibiotic treatment duration in patients with sepsis in the ICU.

Specific Aims

1. To show that implementation of a procalcitonin-guided antibiotics stewardship algorithm may result in shortened antibiotics course in ICU sepsis patients
2. To show that implementation of a procalcitonin-guided antibiotics stewardship algorithm may not result in inferior outcome as compared to conventional therapy

ELIGIBILITY:
Inclusion Criteria:

* All patients with laboratory- or image-confirmed severe infection at admission or during stay in ICU will be eligible for inclusion.

Definition of laboratory- or image-confirmed severe infection:

1. Two or more of four Signs of Inflammation

   * Temperature > 38.3℃ or < 36℃
   * Heart rate > 90 beats/min
   * Respiratory rate > 20 breaths/min or PaCO2 < 32 mmHg
   * WBC > 12,000 cells/mm3, < 4000 cells/mm3, or > 10% bands
2. Initial Procalcitonin > 0.5 ng/mL
3. Presence of either laboratory or image evidence of infection

Laboratory evidence:

Sign of inflammation in urine, CSF, ascites, pleural effusion or local abscess

Image evidence:

Compatible findings on Chest X ray、ultrasound、CT、or MR image

Exclusion Criteria:

* Age less than 20 years
* Known pregnancy
* Presence of DNR order
* Expected ICU stay less than 3 days
* Neutropenia (ANC count < 500/mm3)
* Specific infections for which long-term antibiotic treatment is strongly recommended: lung abscess or empyema, bacterial meningitis, osteomyelitis, infective endocarditis, local abscess, mediastinitis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1700 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Average antibiotics duration | 28 days
28-day mortality rate | 28 days
  Safety endpoints

SECONDARY OUTCOMES:
Proportion of antibiotics use in both arms | 28 days
Length of ICU stay | 90 days
Recurrence of fever within 72 hours of antibiotics discontinuation | 28 days
APACHE-II score or SOFA score | 28 days
Reinfection between 72-hours and 28 days post antibiotics discontinuation | 28 days
90-day all-cause mortality | 90 days
90-day infection related readmission rate | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Lee, MD, MSc, Principal Investigator — National Taiwan University Hospital
Locations (8):
- China (6):
  - Department of Critical Care Medicine, The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Department of Critical Care Medicine, The 301 People Liberation Army General Hospital, Beijing
  - Emergency Department, Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Emergency Department, Ruijin Hospital, Jiaotong University, School of Medicine, Shanghai
  - Emergency Department, Xinhua Hospital, Jiaotong University School of Medicine, Shanghai
  - Department of Critical Care Medicine, The General Hospital of Tianjin Medical University, Tianjin
- Department of Pathology, Princess Margaret Hospita, Lai Chi Kok, Hong Kong
- Department of Emergency, National Taiwan University Hospital, Taipei, Taiwan